CLINICAL TRIAL: NCT05089773
Title: Outcomes of Transposition of the Great Arteries After Arterial Switch Operation: a Dual-center Study
Brief Title: Outcomes of Transposition of the Great Arteries After Arterial Switch Operation
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TGA-CTS
Record Dates: First submitted 2021-03-10; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-03

CONDITIONS: Transposition of Great Vessels; Outcome, Fatal
Keywords: arterial switch operation; late referral; transposition of the great arteries
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: The only group in this retrospective study includes patients diagnosed with transposition of the great arteries receiving arterial switch operation in children's hospital of fudan university and shanghai children's medical center.
  Interventions: Procedure: The arterial switch operation

INTERVENTIONS:
Procedure: The arterial switch operation — The ASO is a procedure that emerged as an anatomically as well as physiologically appropriate solution to the transposition of the great arteries. The aorta and pulmonary artery are detached from their native roots and reattached to the opposite root; thus, the pulmonary root becomes the neo-aorta, and the aortic root becomes the neo-pulmonary artery.
  The coronary arteries are transplanted from the aorta/neo-pulmonary artery to the pulmonary artery/neo-aorta.

SUMMARY:
Transposition of the great arteries (TGA) is a complex cyanotic congenital heart disease and patients suffer from a high mortality rate within one year of age without appropriate management. The therapeutic effect of arterial switch operation (ASO) is satisfactory with low surgery mortality of 2-5%, and thus, has become the treatment of choice for surgical correction of d-TGA. Outcomes of ASO in TGA in china are rare. This is a retrospective study reporting the outcomes of ASO in TGA.

DETAILED DESCRIPTION:
Transposition of the Great Arteries (TGA) is a relatively rare congenital heart disease and surgical treatment in China was developed in recent 20 years. The outcomes of arterial switch operation (ASO) in TGA in China have not been reported before. This study was designed to offer the experience of surgical treatment of TGA in two major pediatric heart centers affiliated in national children's medical center in China. In this retrospective study, a total of 1281 patients diagnosed with TGA received ASO treatment in Fudan Children's Hospital and Shanghai Children's Medical Center were recruited. Medical records and follow-up data of patients were complete. Patient characteristics and clinical data were obtained through review of the medical records, preoperative echocardiography and cardiac catheterization data, operative notes, and follow up reports. Description of the anatomy was confirmed on the preoperative echocardiogram, with clarification from the operative note as needed. Anatomy of the coronary arteries were collected based on the surgical notes. Perioperative data included aorta cross clamping time, cardiopulmonary bypass time and the application of Lecompete maneuver.

Early postoperative complications are defined as delayed sternal closure, active bleeding after surgery, pulmonary artery stenosis, coronary artery re-transplantation, residual ventricular septal defect with significant shunt, atrioventricular block, extracorporeal membrane oxygenation support, cardiac arrest, necrotizing enterocolitis and diaphragmatic eventration. Hospital death was defined as death occurred before discharge.

Follow-up results included echocardiography, cardiac CTA, cardiac catheterization, and angiography. Echocardiographic assessment included color, continuous wave, and pulse wave Doppler date for all valves. Peak pressure gradient of 20mmHg was considered to be stenotic for neoaortic and pulmonary valve. Redo-procedure was defined as any kind of cardiovascular intervention after the ASO procedure including surgery or catheter-based procedure. The indication for reintervention of pulmonary or suprapulmonary stenosis was peak pressure gradient over 40mmHg. Pressure gradient across the LVOT or aortic valve over 50 mmHg was the indication for reintervention. Late death was defined as death occurred during follow up.

Relationships between preoperative and perioperative factors and hospital mortality were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with the great arteries receiving the arterial switch operation in children's hospital of Fudan university and Shanghai children's medical center from January 2000 to March 2020.

Exclusion Criteria:

* NA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with the great arteries receiving the arterial switch operation in children's hospital of Fudan university and Shanghai children's medical center from January 2000 to March 2020, regardless of the age, sex, and the anatomy.
Sampling Method: Non-Probability Sample
Enrollment: 1281 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
hospital mortality | within 1 month after ASO
  death occurred within the hospital
late death | after 1 month after ASO
  death occurred after discharge
redo operation | through study completion, an average of 10 year
  reintervention after the ASO procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bing Jia, MD, PhD, Study Chair — Children's Hospital of Fudan University
Locations (2):
- China (2):
  - Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's medical center, Shanghai

IPD SHARING:
Plan to Share IPD: No